CLINICAL TRIAL: NCT06484933
Title: Assessing Risk Management in Primary Care Teams
Brief Title: Risk Management in Primary Care
Acronym: eGERISSEP
Status: Not yet recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL24_0010
Record Dates: First submitted 2024-06-10; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Primary Care
Keywords: Primary care; Risk management; Teamwork

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthcare professionals and users of primary care: Health professionals and users of primary care will be asked during focus groups on the definition of the professional team in primary care and on the risk management procedures put in place in primary care organisations.
  Interventions: Behavioral: Focus groups of health professionals and users of primary care

INTERVENTIONS:
Behavioral: Focus groups of health professionals and users of primary care — 2 phases of Focus Group will be organized :
  * the participants of the first 4 Focus Groups will propose an operational definition of the notion of a professional team in primary care (validation by consensus based on the definitions in the literature)
  * 12 subsequent Focus Groups will be organized in 12 primary care teams to describe the ways in which risks are managed in primary care

SUMMARY:
The proposed research is a prospective, non-comparative study based on a qualitative method, comprising a literature review followed by 2 successive series of Focus Groups with users and healthcare professionals of primary care in the French AURA region. The 2 Focus Group phases will make it possible to :

* propose an operational definition of the notion of a professional team in primary care (validation by consensus between the participants of the first 4 Focus Groups based on the definitions in the literature)
* describe the ways in which risks are managed in primary care teams (qualitative analysis of the contributions made by the participants in the next 12 Focus Groups organized in 12 primary care teams)

ELIGIBILITY:
Inclusion Criteria:

Healthcare professional

* Healthcare professional over 18 years of age, registered with the professional association on which he/she depends and holding an RPPS identification number with care activity as part of a coordinated practice, within a legally formalised care team working on a territorial health project, or care activity within a care team that is not legally formalized but defined as an entity bringing together ≥ 4 different professionals to care for the same patient.
* Most care provided on an outpatient basis
* Care activity in the AURA region
* Agreement to participate in the focus group Users
* Any user of the healthcare system over the age of 18
* Consulting a healthcare professional from a team included in the research
* Agreement to participate in the focus group

Exclusion Criteria:

Healthcare professional

* Primary care healthcare professional with a specific exclusive practice that does not form part of the overall management of a patient (e.g. homeopathy, mesotherapy, acupuncture, etc.) Users
* Persons deprived of their liberty by a judicial or administrative decision
* Adults under legal protection (guardianship, curatorship)
* Persons not affiliated to a social security scheme or beneficiaries of a similar scheme

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care organizations in France
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07-05 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Operational definition of the notion of a professional team in primary care in the France, by means of focus groups and validation by consensus. | up to 23 months
  This definition will be based on data from a literature review adapted to the context of French primary care and the practices/experience of professionals and users by means of focus groups including professionals and users from the primary care teams.

CONTACTS AND LOCATIONS:
Locations (1):
- Cabinet Medical, Oullins, France